CLINICAL TRIAL: NCT02531516
Title: ATLAS: A Randomized, Double-blind, Placebo-controlled Phase 3 Study of JNJ-56021927 in Subjects With High-risk, Localized or Locally Advanced Prostate Cancer Receiving Treatment With Primary Radiation Therapy
Brief Title: An Efficacy and Safety Study of JNJ-56021927 (Apalutamide) in High-risk Prostate Cancer Subjects Receiving Primary Radiation Therapy: ATLAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR106935; 56021927PCR3003 (Other: Janssen Research & Development, LLC); 2015-003007-38 (EudraCT Number); 2023-505246-26-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2015-08-21; First posted 2015-08-24 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic neoplasms; Prostate Cancer; High-Risk prostate cancer; JNJ-56021927; Apalutamide; ATLAS; Radiation; Long-term hormone therapy; Localized or locally advanced prostate cancer; Janssen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; bicalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Apalutamide (Experimental): Participants will receive apalutamide (240 mg), by mouth, once daily for overall 30 months, plus bicalutamide placebo, by mouth, once daily, for four months from randomization. All participants are treated with gonadotropin releasing hormone (GnRH) agonist for 30 months from randomization and radiation therapy to the prostate started at about 8 weeks after randomization.
  Interventions: Drug: Apalutamide; Drug: Bicalutamide Placebo; Drug: GnRH (agonist); Radiation: 74-80 Grays (units of radiation)
- Control group (Active Comparator): Participants will receive apalutamide placebo, by mouth, once daily for overall 30 months, plus bicalutamide (50 mg), by mouth, once daily, for four months from randomization. All participants are treated with gonadotropin releasing hormone (GnRH) agonist for 30 months from randomization and radiation therapy to the prostate started at about 8 weeks after randomization.
  Interventions: Drug: Bicalutamide; Drug: Apalutamide Placebo; Drug: GnRH (agonist); Radiation: 74-80 Grays (units of radiation)

INTERVENTIONS:
Drug: Apalutamide
  Arms: Apalutamide
Drug: Bicalutamide
  Arms: Control group
Drug: Bicalutamide Placebo
  Arms: Apalutamide
Drug: Apalutamide Placebo
  Arms: Control group
Drug: GnRH (agonist)
Radiation: 74-80 Grays (units of radiation)

SUMMARY:
The purpose of this study is to determine if apalutamide plus gonadotropin releasing hormone (GnRH) agonist in participants with high-risk, localized or locally advanced prostate cancer receiving primary radiation therapy (RT) results in an improvement of metastasis-free survival (MFS) based on conventional imaging assessed by blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Indicated and planned to receive primary radiation therapy for prostate cancer
* Histologically confirmed adenocarcinoma of an intact prostate, and 1 of the following at diagnosis: 1) Gleason score >=8 and >=cT2c, 2) Gleason score 7, PSA >=20 nanogram per milliliters (ng/mL), and >=cT2c
* Charlson index (CCI) <=3
* An Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) grade of 0 or 1
* Adequate organ function: (1) aspartate aminotransferase (AST), alanine aminotransferase (ALT), within normal limits (WNL), (2) serum creatinine less than (<) 1.5 milligram/deciliter (mg/dL) (<133 micromoles/Liter [mcmol/L]), (3) platelets greater than or equal to (>=)140,000/microLiter (mcL), independent of transfusion and/or growth factors within 3 months prior to randomization, (4) Hemoglobin >= 12.0 gram/deciliter (g/dL) (7.4 millimloes [mmol], independent of transfusion and/or growth factors within 3 months prior to randomization
* Participants who are sexually active (even men with vasectomies) and willing to use a condom and agree not to donate sperm during the trial
* Signed, written, informed consent
* Be able to swallow whole study drug tablets

Exclusion Criteria: -

* Presence of distant metastasis, (clinical stage M1). Isolated pelvic nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion. Diagnosis of distant metastasis (clinical M stage; M0 versus M1a, M1b, M1c) and pelvic nodal disease (clinical N stage; N1 versus N0) will be assessed by central radiological review. Patients are considered eligible only if the central radiological review confirms clinical stage M0
* Prior treatment with gonadotropin releasing hormone (GnRH) analogue or anti-androgen or both for >3 months prior to randomization
* Bilateral orchiectomy
* History of pelvic radiation
* Prior systemic (example [e.g.], chemotherapy) or local (e.g. radical prostatectomy, cryotherapy) treatment for prostate cancer
* History of seizure or any condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness <= 1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect)
* Prior treatment with enzalutamide, abiraterone acetate, orteronel, galeterone, ketoconazole, aminoglutethimide, estrogens, megestrol acetate, and progestational agents (including cyproterone acetate) for prostate cancer
* Prior treatment with radiopharmaceutical agents (e.g., strontium-89) or immunotherapy (e.g., sipuleucel-T) for prostate cancer
* Prior treatment with systemic glucocorticoids ≤4 weeks prior to randomization or is expected to require long-term use of corticosteroids during the study
* Use of 5-alpha reductase inhibitors (e.g., dutasteride, finasteride) <=4 weeks prior to randomization
* Use of any investigational agent <=4 weeks prior to randomization
* Current chronic use of opioid analgesics for >=3 weeks for oral or >= 7 days for non-oral formulations
* Major surgery <=4 weeks prior to randomization
* Current or prior treatment with anti-epileptic medications for the treatment of seizures
* Gastrointestinal conditions affecting absorption
* Known or suspected contraindications or hypersensitivity to apalutamide, bicalutamide or GnRH agonists or any of the components of the formulations
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Metastasis-Free Survival (MFS) | 108 Months
  MFS is defined as the time from randomization to the date of the first occurrence of radiographic bone or soft tissue distant metastasis based on conventional imaging assessed by blinded independent central review (BICR), histopathologic diagnosis of distant metastasis, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Event-Free Survival (EFS) Based on Conventional Imaging Assessed By BICR | 108 Months
  EFS is defined as the time from randomization to the date of the first occurrence of prostate specific antigen (PSA) failure by the Phoenix definition, local or regional disease recurrence based on conventional imaging assessed by BICR or histopathologic diagnosis, distant metastasis based on conventional imaging assessed by BICR or histopathologic diagnosis, or death.
Time to PSA Progression | 108 Months
  Time to PSA progression is defined as the time from randomization to the date of PSA nadir plus (+) 0.5 nanograms per milliliter (ng/mL) and rising.
MFS Based on Conventional Imaging or Prostate-Specific Membrane Antigen (PSMA)-Positron Emission Tomography (PET) Imaging Assessed by BICR | 108 Months
  MFS is defined as the time from randomization to the date of the first occurrence of radiographic bone or soft tissue distant metastasis based on conventional imaging assessed by BICR or PSMA-PET imaging assessed by BICR, histopathologic diagnosis of distant metastasis, or death from any cause, whichever occurs first.
No Evidence of Disease (NED) Based on Conventional Imaging or PSMA PET Imaging Assessed by BICR | 108 Months
  NED is defined as: alive; no PSA progression; no distant metastasis based on conventional imaging assessed by BICR or PSMA-PET imaging assessed by BICR or histopathologic diagnosis; no local or regional recurrence based on conventional imaging assessed by BICR or PSMA-PET imaging assessed by BICR, or histopathologic diagnosis; no subsequent therapy for prostate cancer; testosterone recovery to age-related pre-androgen deprivation therapy (pre-ADT)/baseline or greater than (>) 200 nanogram per deciliter (ng/dL).
Overall Survival (OS) | 108 Months
  OS is defined as the time from randomization to date of death from any cause.
Time to Distant Metastasis Based on Conventional Imaging Assessed by BICR | 108 Months
  Time to distant metastasis is defined as the time from randomization to the date of the first occurrence of radiographic or pathological bone or soft tissue distant metastasis based on conventional imaging assessed by BICR or histopathologic diagnosis of distant metastasis.
EFS Based on Conventional Imaging or PSMA-PET Imaging Assessed by BICR | 108 Months
  EFS is defined as the time from randomization to the date of the first occurrence of PSA failure by the Phoenix definition, local or regional disease recurrence based on conventional imaging assessed by BICR or PSMA-PET imaging assessed by BICR or histopathologic diagnosis, distant metastasis based on conventional imaging assessed by BICR or PSMA-PET imaging assessed by BICR or histopathologic diagnosis, or death.
Time to Next Local or Systemic Treatment | 108 Months
  Time to next local or systemic treatment is defined as the time from randomization to the first subsequent therapy, including re-initiation of androgen deprivation therapy (ADT) and local treatments for local-regional recurrence or distant metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Aragon Pharmaceuticals, Inc. Clinical Trial, Study Director — Aragon Pharmaceuticals, Inc.
Locations (262):
- United States (60):
  - Homewood, Alabama
  - Chandler, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Bakersfield, California
  - Los Angeles, California
  - Orange, California
  - San Bernardino, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Denver, Colorado
  - Middlebury, Connecticut
  - Bradenton, Florida
  - Daytona Beach, Florida
  - Fort Myers, Florida
  - Hialeah, Florida
  - Lakewood Rch, Florida
  - Naples, Florida
  - Plantation, Florida
  - Meridian, Idaho
  - Evergreen Park, Illinois
  - Harvey, Illinois
  - Jeffersonville, Indiana
  - Wichita, Kansas
  - Ashland, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - St Louis, Missouri
  - Morristown, New Jersey
  - Albany, New York
  - Brooklyn, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Cary, North Carolina
  - Raleigh, North Carolina
  - Portland, Oregon
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - East Greenwich, Rhode Island
  - Charleston, South Carolina
  - Myrtle Beach, South Carolina
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Virginia Beach, Virginia
  - Burien, Washington
  - Spokane, Washington
  - Morgantown, West Virginia
- Argentina (6):
  - Buenos Aires
  - C.a.b.a.
  - Caba
  - Pergamino
  - Rosario
  - San Salvador de Jujuy
- Belgium (11):
  - Aalst
  - Antwerp
  - Bonheiden
  - Brussels
  - Haine-St-Paul
  - Leuven
  - Liège
  - Namur
  - Roeselare
  - Sint-Niklaas
  - Turnhout
- Brazil (16):
  - Barretos
  - Belo Horizonte
  - Campinas
  - Curitiba
  - Florianópolis
  - Goiânia
  - Ijuí
  - Natal
  - Porto Alegre
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - Santo André
  - São José do Rio Preto
  - São Paulo
  - Sorocaba
- Canada (12):
  - Calgary, Alberta
  - Surrey, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Gatineau, Quebec
  - Laval, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Sherbrooke, Quebec
- China (11):
  - Beijing
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Nanchang
  - Nanjing
  - Ningbo
  - Shanghai
  - Wuhan
  - Xi'an
- Czechia (8):
  - Hradec Králove
  - Liberec
  - Nový Jicin
  - Olomouc
  - Opava
  - Pardubice
  - Prague
  - Zlín
- France (28):
  - Amiens
  - Angers
  - Avignon
  - Bayonne
  - Besançon
  - Bordeaux
  - Brest
  - Dijon
  - Évry-Courcouronnes
  - Hyères
  - La Tronche
  - Le Mans
  - Lille
  - Marseille
  - Marseilli
  - Montpellier
  - Neuilly-sur-Seine
  - Paris
  - Ris-Orangis
  - Saint-Brieuc
  - Saint-Herblain
  - Saint-Mandé
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy
  - Villejuif
- Germany (10):
  - Braunschweig
  - Chemnitz
  - Dessau
  - Frankfurt
  - Gronau
  - Jena
  - Münster
  - Nürtingen
  - Ulm
  - Weiden/Opf
- Israel (8):
  - Beer Yaakov
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Malaysia (4):
  - George Town
  - Kuala Lumpur
  - Kuching
  - Putrajaya
- Mexico (6):
  - Culiacán
  - Guadalajara
  - León
  - México
  - Morelia
  - Zapopan
- Netherlands (5):
  - Alkmaar
  - Amsterdam
  - Nijmegen
  - Rotterdam
  - The Hague
- Poland (9):
  - Bialystok
  - Bydgoszcz
  - Gdynia
  - Gliwice
  - Kielce
  - Lodz
  - Olsztyn
  - Poznan
  - Wałbrzych
- Romania (9):
  - Bucharest
  - Cluj-Napoca
  - Floreşti
  - Iași
  - Otopeni
  - Ploieşti
  - Sibiu
  - Târgu Mureş
  - Timișoara
- Russia (15):
  - Barnaul
  - Ivanovo
  - Moscow
  - Nizhny Novgorod
  - Obninsk
  - Omsk
  - Pyatigorsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Saransk
  - Tambov
  - Tyumen
  - Ufa
  - Vologda
- South Korea (4):
  - Daegu
  - Gyeonggi-do
  - Jeollanam-do
  - Seoul
- Spain (10):
  - Barakaldo
  - Barcelona
  - Castellon
  - L'Hospitalet de Llobregat
  - Las Palmas de Gran Canaria
  - Madrid
  - Málaga
  - Reus
  - Santiago de Compostela
  - Seville
- Sweden (3):
  - Örebro
  - Stockholm
  - Umeå
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
- Turkey (Türkiye) (7):
  - Adana
  - Ankara
  - Edirne
  - Istanbul
  - Izmir
  - Kayseri
  - Kocaeli
- Ukraine (4):
  - Dnipro
  - Khakhiv
  - Kyiv
  - Lviv
- United Kingdom (11):
  - Aberdeen
  - Birmingham
  - Bristol
  - Derby
  - Glasgow
  - Oxford
  - Plymouth
  - Preston
  - Sheffield
  - Sutton
  - Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poterala JE, Wisinski KB. Abbreviated endocrine therapy duration for low estrogen receptor-positive breast cancer: The counter to extended endocrine therapy. Cancer. 2022 May 1;128(9):1724-1726. doi: 10.1002/cncr.34158. Epub 2022 Feb 25. No abstract available. PMID 35213039